CLINICAL TRIAL: NCT04457089
Title: Statin Therapy to Reduce Progression in Women With Platinum Sensitive Ovarian Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Marc Goodman (Other)
Responsible Party: Sponsor-Investigator, Marc Goodman, Oncologist, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2020-03-Rimel-STOV
Record Dates: First submitted 2020-06-25; First posted 2020-07-07 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Recurrent Ovarian Cancer; Platinum-sensitive Ovarian Cancer
Keywords: simvastatin
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Simvastatin (Experimental)
  Interventions: Drug: Simvastatin 40mg

INTERVENTIONS:
Drug: Simvastatin 40mg — Simvastatin 40mg by mouth nightly for approximately 6 months during treatment with carboplatin and liposomal doxorubicin
  Other Names: Zocor

SUMMARY:
This is a single arm pilot trial to evaluate the feasibility of using a simvastatin intervention, and to evaluate its effects on cancer progression, among 20 patients with platinum-sensitive ovarian cancer, treated with carboplatin and liposomal doxorubicin at Cedars-Sinai Medical Center.

DETAILED DESCRIPTION:
This is a pilot study of statin therapy to examine the feasibility of simvastatin use to reduce disease progression in 20 patients with platinum-sensitive ovarian cancer at Cedars-Sinai Medical Center. This study will focus on patients with recurrent platinum sensitive ovarian cancer to increase the likelihood that this population will experience recurrent disease during the 6-month intervention and follow-up. In addition, this population of patients has a narrow range of standard of care carboplatin doublet combinations that are prescribed, enabling the investigators to create a more homogenous study population. Given their high risk of developing recurrent disease, women with platinum sensitive ovarian cancer, have the potential to derive the maximum benefit from an intervention that could delay disease progression and enhance survival.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent platinum sensitive ovarian cancer, all histologies (serous, endometrioid, mucinous, clear cell). Platinum sensitivity defined as ≥ 6 months since last platinum treatment.
* No contraindication to carboplatin and/or liposomal doxorubicin or simvastatin.

Exclusion Criteria:

* Prior or current use of any statin medication
* Current systemic use of medications known to interact with statins
* Current use of any other investigational agents
* Liver disease, active cirrhosis
* Uncontrolled intercurrent illness
* History of chronic myopathy
* Prior cancer other than ovarian cancer or non-melanomatous skin cancers
* Known active infection with HIV
* Current excessive alcohol consumption (average alcohol consumption of more than 5 drinks per day)
* Prior exposure to doxorubicin or liposomal doxorubicin
* Hemoglobin A1C >8.0%

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-05-12 (Actual)

PRIMARY OUTCOMES:
Completion of the simvastatin intervention with at least 85% compliance | From Cycle 1 Day 1 until Cycle 6 Day 28 (each cycle is 28 days)
  Percentage of patients who complete the simvastatin intervention with at least 85% compliance during Carboplatin and Doxil chemotherapy.

SECONDARY OUTCOMES:
Response by CA125 | From baseline until 12 months
  Change in serum level of CA125
Progression-free survival | From baseline until 12 months
  Duration until disease progression or death

CONTACTS AND LOCATIONS:
Overall Officials: Bobbie Jo Rimel, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No